CLINICAL TRIAL: NCT03785886
Title: Intervention Effects and Safety Evaluation of Different Exercise Training Programs on Hypertension and Hypertension Complicated With Diabetes
Brief Title: Effects of Different Training Programs in Chronic Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Sport University (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016YFC1300202
Record Dates: First submitted 2018-11-29; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Hypertension; Hypertension Complicated With Type 2 Diabetes; Walking; Chinese Square Dancing
Keywords: hypertension; hypertension complicated with type diabetes; walking; Chinese square dancing
MeSH Terms: conditions — Hypertension | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Walking group (Experimental): The study is a randomized 3-month community-based exercise intervention with a control group and 2 different exercise groups: walking group and Chinese square dancing group.
  Eighteen communities will be selected in Beijing, and they will be age matched and randomly grouped into walking, Chinese square dancing and control groups. Each community will include twenty subjects (ten patients with hypertension and ten patients with hypertension complicated with type 2 diabetes) aged 40-69 years.
  Interventions: Behavioral: Walking group
- Chinese Square Dancing group (Experimental): The study is a randomized 3-month community-based exercise intervention with a control group and 2 different exercise groups: walking group and Chinese square dancing group.
  Eighteen communities will be selected in Beijing, and they will be age matched and randomly grouped into walking, Chinese square dancing and control groups. Each community will include twenty subjects (ten patients with hypertension and ten patients with hypertension complicated with type 2 diabetes) aged 40-69 years.
  Interventions: Behavioral: Chinese square dancing group
- Control group (Experimental): The study is a randomized 3-month community-based exercise intervention with a control group and 2 different exercise groups: walking group and Chinese square dancing group.
  Eighteen communities will be selected in Beijing, and they will be age matched and randomly grouped into walking, Chinese square dancing and control groups. Each community will include twenty subjects (ten patients with hypertension and ten patients with hypertension complicated with type 2 diabetes) aged 40-69 years.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Walking group — Subjects in this group perform exercise consisting of walking for 30 - 60 min at 40% - 60% HRR intensity 3-5 d•wk-1 for 3 months . Each training includes 5 min warm-up and 5 min cool-down, and the exercise should start after meals for 1 hour . Heart rate is monitored by sports bracelet . Subjects using β-blockers will not use heart rate to monitor exercise intensity , but RPE scores . And RPE( Borg scale) scores are ranged from 11-13.
  Arms: Walking group
Behavioral: Chinese square dancing group — Chinese square dances have been selected from 24 sets of square dances jointly launched in 2015 and 2017. According to the age and physical health status of the subjects, six dance pieces of are selected as the repertoires of the intervention in this study.
  Subjects in this group perform exercise consisting of Chinese square dances for 30-60 min at 40% - 60% HRR intensity 3-5 d•wk-1 for 3 months. Each training includes 5 min warm-up and 5 min cool-down , and the exercise should start after meals for 1 hour. Make the subjects step for 30 s to 1 min between each track to adjust the heart rate. Heart rate is monitored by sports bracelet. Subjects using β-blockers will not use heart rate to monitor exercise intensity, but RPE scores. And RPE( Borg scale) scores are ranged from 11-13.
  Arms: Chinese Square Dancing group
Behavioral: Control group — Walking group , Chinese square dancing group and control group are given the same health education brochures or health education lectures once a month . Specific contents of the brochure or lecture include : type 2 diabetes , hypertension related medical knowledge and the significance of intervention treatment ; prevention of type 2 diabetes , hypertension nutrition and exercise recommendations ; basic knowledge of scientific exercise and its matters needing attention .
  Arms: Control group

SUMMARY:
The study is a randomized 3-month community-based exercise intervention with a control group and 2 different exercise groups: walking group and Chinese square dancing group.Eighteen communities will be selected in Beijing, and they will be age matched and randomly grouped into walking, Chinese square dancing and control groups. Each community will include twenty subjects (ten patients with hypertension and ten patients with hypertension complicated with diabetes) aged 40-69 years. All exercise sessions will be supervised and subject's exercise implementation process will be managed with intelligent equipment. The purpose of the study is to evaluate the effectiveness and safety of different training programs.

The demographics data, physical activity questionnaires, blood pressure, blood glucose, blood lipids, height, weight and physical fitness （cardiorespiratory fitness，muscle strength, muscle endurance, flexibility, body composition） will be measured before and after 3-month exercise training .The adverse reactions in the implementation of the interventions will be recorded. The primary outcomes are blood pressure and blood glucose.

DETAILED DESCRIPTION:
The global burden of disease study shows that unreasonable diets and physical inactivity are the largest health risks facing the world today. In recent years, foreign and domestic scholars have gradually introduced the concept of " Exercise is Medicine " guide the the public exercise scientifically. However, under the special cultural background of China, it is urgent to answer how to help the public to realize reasonable scientific exercise, how to choose the popular exercise mode and whether the exercise mode is scientific and effective.

Previous meta-analysis studies on the improvement of blood pressure and blood glucose by walking have been published, but few studies on Chinese square dancing have been conducted. Previous studies on whether Chinese square dancing was scientific and effective were mostly small sample population studies carried out by Chinese scholars. The research results were of large heterogeneity, and the research design lacked reasonable consideration.

This study intends to select two common exercise mode for scientific evaluation, one is walking and the other is Chinese square dancing. The purpose of this study is to evaluate the efficacy and safety of two common types of exercise (walking and Chinese square dancing) in Chinese patients with hypertension and patients with hypertension complicated with diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. 40-69 years of age
2. Meet any one of the two conditions:

   2.1 Hypertension: diagnosed with hypertension, systolic blood pressure is 130-159 mmHg, take no antihypertensive drug or no more than 2 kinds of antihypertensive drugs

   2.2 Hypertension complicated with diabetes: diagnosed with hypertension and type 2 diabetes, systolic blood pressure is 130-159 mmHg and the fasting blood glucose in the past 2 weeks was 5.6-16.7 mmol/L (13.8-16.7 mmol/L was negative for urinary ketone) , take no more than 4 kinds of antihypertensive and hypoglycemic drugs
3. Maintain the current state of medication for the next 3 months
4. Lived in the current community in the past six months
5. Have no intention of moving out for the next three months
6. Have no regular exercise habit (moderate intensity activity less than 3 times a week, less than 30 minutes each time or 30 minutes cumulative), at least exercise 3 days a week
7. Sign informed consent

Exclusion Criteria:

1. Manual works(such as farmers, couriers, athletes and workers, who rely on physical activity to make a living)
2. Physical disability that prevents patients from walking or Chinese square dancing
3. Currently enrolled in another lifestyle intervention trial(interventions such as nutrition, psychology, exercise and health education)
4. Pregnant or planning to become pregnant
5. BMI(body mass index)≥35 kg/m2
6. Answers to questions 2, 3 and 6 of the questionnaire in 2014PAR-Q+ are "yes"
7. Cardio-cerebrovascular events have occurred in the past 6 months(heart disease diagnosed by doctors, such as coronary heart disease, hypertensive heart disease, acute myocarditis, pulmonary heart disease, etc.)
8. Fasting blood glucose of diabetic patients is 13.8-16.7 mmol/L and urinary ketone is positive
9. Severe complications of diabetes affecting exercise , such as foot, eye disease and renal insufficiency
10. Complicated with other serious chronic diseases such as asthma, malignant tumor, chronic heart failure, severe depression or other mental disorders

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Systolic Blood Pressure at 3 months | Before and after interventions（3 months)
  To evaluate the effect of walking and Chinese square dancing on systolic blood pressure in hypertensive patients and patients with hypertension complicated with type 2 diabetes.
Change from Baseline Fasting Blood Glucose at 3 months | Before and after interventions（3 months）
  To evaluate the effect of walking and Chinese square dancing on fasting blood glucose in hypertensive patients and patients with hypertension complicated with type 2 diabetes.

SECONDARY OUTCOMES:
Change from Cardiorespiratory Fitness at 3 months | Before and after interventions（3 months）
  To evaluate the effect of walking and Chinese square dancing on cardiorespiratory fitness in hypertensive patients and patients with hypertension complicated with type 2 diabetes. Cardiorespiratory fitness (2 minutes high knee lift) is in heart beats per minute.
Change from Muscle Strength at 3 months | Before and after interventions（3 months）
  To evaluate the effect of walking and Chinese square dancing on muscle strength in hypertensive patients and patients with hypertension complicated with type 2 diabetes. Muscle strength (grip strength) is in kilograms.
Change from Muscle Endurance at 3 months | Before and after interventions（3 months）
  To evaluate the effect of walking and Chinese square dancing on muscle endurance in hypertensive patients and patients with hypertension complicated with type 2 diabetes. Muscle endurance (40-59 yrs: push-ups(male) or sit-ups(female), 60-69 yrs: 30-second chair stand test and 30-second arm curl test) is in numbers.
Change from Flexibility at 3 months | Before and after interventions（3 months）
  To evaluate the effect of walking and Chinese square dancing on flexibility in hypertensive patients and patients with hypertension complicated with type 2 diabetes. Flexibility (40-59 yrs :reach test, 60-69 yrs : chair sit-and-reach test) is in centimeters.
Change from Balance at 3 months | Before and after interventions（3 months）
  To evaluate the effect of walking and Chinese square dancing on balance in hypertensive patients and patients with hypertension complicated with type 2 diabetes. Balance (standing on one leg with eyes closed) is in seconds.
Change from Body Composition at 3 months | Before and after interventions（3 months）
  To evaluate the effect of walking and Chinese square dancing on body composition in hypertensive patients and patients with hypertension complicated with type 2 diabetes. Body composition (bioelectrical impedance ) is in percentage of weight.
Time and Frequency of Adverse Reactions and Serious Adverse Events through the study completion | Every day during the interventions until the end of the study（3 months）
  This study will collect the following safety information and record it in the CRF, including: research-related adverse reactions and serious adverse events. The relevant definitions and procedures are as follows.
  The adverse effects of exercise include: cardiovascular and cerebrovascular diseases, aggravation of complications associated with diabetes/hypertension, and sports injuries. Severe adverse events (SAEs) are defined as conditions that result in any of the following outcomes after exercise intervention: death, life-threatening, hospitalization, permanent or significant disability, dysfunction.
  If a SAE occurs during the course of the study, the investigator should immediately take appropriate treatment on the subject and terminate the trial. Adverse reactions are asked daily by the researcher. In the event of an adverse reaction, the investigator is required to record the following in the CRF: the time, severity, end time, measures taken, and outcome of the adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengzhen Wang, Doctor, Study Director — Beijing Sport University
Locations (1):
- School of Sport Medicine and Rehabilitation，Beijing Sport University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided